CLINICAL TRIAL: NCT06724237
Title: A Randomized Phase III Study to Evaluate Benefits of Autologous Stem Cell Transplant in Patients With Peripheral T Cell Lymphoma That Achieved a First Complete Remission (CR1) Following Induction Therapy (PTCL-STAT)
Brief Title: Testing Whether High Dose Chemotherapy and Infusion of the Patients' Own Stem Cells Improves Survival in Patients With Peripheral T-cell Lymphoma Who Achieved a Complete Response at the End of the Initial Chemotherapy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA4232; NCI-2024-06604 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA4232 (Other: ECOG-ACRIN Cancer Research Group); EA4232 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-11-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-08

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Negative; Follicular Helper T-Cell Lymphoma; Follicular Helper T-Cell Lymphoma, Angioimmunoblastic-Type; Peripheral T-Cell Lymphoma, Not Otherwise Specified
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell | interventions — Stem Cell Transplantation; Practice Guidelines as Topic; Standard of Care; Specimen Handling; Biopsy; Drug Therapy; Leukapheresis; Magnetic Resonance Spectroscopy; Hematopoietic Stem Cell Mobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (observation) (Active Comparator): Patients receive standard of care observation on study. Patients also undergo blood sample collection and optional bone marrow aspiration and biopsy on study, and CT or PET/CT throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography
- Arm II (high dose chemotherapy and ASCT) (Experimental): Patients receive stem cell mobilization and then undergo leukapheresis per standard of care. Patients also receive high dose chemotherapy followed by ASCT per standard of care. Additionally, patients undergo blood sample collection and optional bone marrow aspiration and biopsy on study, and CT or PET/CT throughout the study.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: High Dose Chemotherapy; Procedure: Leukapheresis; Procedure: Positron Emission Tomography; Drug: Stem Cell Mobilization Therapy

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
  Arms: Arm II (high dose chemotherapy and ASCT)
Other: Best Practice — Receive standard of care observation
  Other Names: standard of care; standard therapy
  Arms: Arm I (observation)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: High Dose Chemotherapy — Receive high dose chemotherapy
  Other Names: high-dose chemotherapy
  Arms: Arm II (high dose chemotherapy and ASCT)
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
  Arms: Arm II (high dose chemotherapy and ASCT)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Stem Cell Mobilization Therapy — Receive stem cell mobilization therapy
  Other Names: Chemomobilization; Hematopoietic Stem Cell Mobilization; Mobilization Therapy; Stem-cell mobilization
  Arms: Arm II (high dose chemotherapy and ASCT)

SUMMARY:
This phase III trial compares the effect of high dose chemotherapy and the patients' own (autologous) stem cells to observation only in patients with peripheral T-cell lymphoma who achieved a complete response after initial chemotherapy. Usual treatment after a complete response may include observation or high dose chemotherapy followed by an autologous stem cell transplant, however, it is not known if a transplant if beneficial. Giving chemotherapy before a stem cell transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. Stem cells removed prior to treatment are then returned to the patient to replace the blood forming cells that were destroyed by the chemotherapy. Giving high dose chemotherapy followed by an autologous stem cell transplant may be more effective compared to observation only in treating patients with peripheral T-cell lymphoma who have achieved a complete response after initial chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate improvement in progression free survival (PFS) in the autologous stem cell transplant (ASCT) arm compared to the observation arm.

SECONDARY OBJECTIVES:

I. To assess difference in overall survival (OS) between the observation and autologous stem cell transplant (ASCT) arm.

II. To evaluate the differences in study intervention benefit for PFS and OS by the randomization stratification factors (histology and choice of induction chemotherapy).

III. To evaluate the cumulative incidence of relapse and mortality between the observational and autologous stem cell transplant (ASCT) arm.

EXPLORATORY OBJECTIVE:

I. To determine the impact of minimal residual disease (MRD) on the benefit of autologous stem cell transplant (ASCT).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care observation on study. Patients also undergo blood sample collection and optional bone marrow aspiration and biopsy on study, and computed tomography (CT) or positron emission tomography (PET)/CT throughout the study.

ARM II: Patients receive stem cell mobilization and then undergo leukapheresis per standard of care. Patients also receive high dose chemotherapy followed by ASCT per standard of care. Additionally, patients undergo blood sample collection and optional bone marrow aspiration and biopsy on study, and CT or PET/CT throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then yearly for up to 7 years for a total of 12 years from the date of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 to 75 years of age
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patient must have histologically proven peripheral T-cell lymphoma (PTCL) in one of the following categories:

  * Anaplastic large cell lymphoma (ALCL) ALK-negative
  * Angioimmunoblastic T-cell lymphoma (AITL)
  * Nodal PTCL with follicular helper T cell (TFH) phenotype
  * Peripheral T-cell lymphoma not otherwise specified (PTCL-NOS)
* Patient must have undergone induction treatment with an anthracycline based chemotherapy.

  * NOTE: Patients who discontinued anthracycline during treatment are eligible as long as they received at least one dose and achieved complete remission
* Patient must have achieved radiologic complete remission following induction therapy as defined by the Lugano criteria with a Deauville score between 1-3 by PET-CT

  * NOTE: There is no central review required. Confirmation of complete remission status is determined by the enrolling institution's review
  * NOTE: If a patient had a positive bone marrow biopsy at the time of initial diagnosis (pre-induction), a repeat biopsy must be completed post induction to confirm complete remission (CR)
* Patient must be eligible for high dose chemotherapy and autologous stem cell transplant (ASCT) per the enrolling institutional guidelines at the transplant center and be ready to proceed with ASCT if randomized to the ASCT arm
* Patient must not have active infection requiring intravenous systemic antimicrobial at time of randomization. Antibiotic prophylaxis is acceptable as long as the dose of the medication has been stable for at least 7 days prior to randomization
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy. A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse during the treatment phase of the study and thereafter according to institutional guidelines
* Absolute neutrophil count (ANC) ≥ 1000/mcL (obtained ≤ 14 days prior to protocol randomization)
* Platelets ≥ 75,000/mcL (obtained ≤ 14 days prior to protocol randomization)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (obtained ≤ 14 days prior to protocol randomization)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3.0 x institutional ULN (obtained ≤ 14 days prior to protocol randomization)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2033-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From study randomization to documented disease progression or death, whichever occurs first, assessed up to 12 years
  Stratified logrank test will be used for the primary analysis of the comparison of PFS between treatment arms. Kaplan-Meier method will be used to visualize and estimate survival function for failure time endpoints. There will be a subgroup analysis for the randomization stratification factors, and other variables measured at baseline.

SECONDARY OUTCOMES:
Overall survival (OS) | From study randomization to death due to any cause, assessed up to 12 years
  Stratified logrank test will be used for the primary analysis of the comparison of OS between treatment arms. Kaplan-Meier method will be used to visualize and estimate survival function for failure time endpoints. There will be a subgroup analysis for the randomization stratification factors, and other variables measured at baseline.
Cumulative incidence of relapse | Up to 12 years
  The cumulative incidence of relapse will be analyzed under the competing risk framework using competing risk regression and competing risk cumulative incidence function plots.
Cumulative incidence of mortality | Up to 12 years
  The cumulative incidence of mortality will be analyzed under the competing risk framework using competing risk regression and competing risk cumulative incidence function plots.

OTHER OUTCOMES:
Proportion of patients with minimal residual disease (MRD) negative result after autologous stem cell transplant (ASCT) in arm B | Up to 12 years
  The proportion of patients with MRD negative results after ASCT will be reported among arm B patients. MRD negative is defined as no lymphoma cell detected.

CONTACTS AND LOCATIONS:
Overall Officials: Nabila N Bennani, Principal Investigator — ECOG-ACRIN Cancer Research Group